CLINICAL TRIAL: NCT01548001
Title: A Randomized, Double-blind Study to Evaluate the Efficacy and Safety of Iguratimod Alone or Iguratimod in Combination With Methotrexate Versus Methotrexate Alone in Patients With Rheumatoid Arthritis
Brief Title: Long-term Efficacy of Iguratimod Alone or Iguratimod in Combination With Methotrexate in Patients With Rheumatoid Arthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM-106
Record Dates: First submitted 2012-03-05; First posted 2012-03-08 (Estimated); Last update posted 2016-02-23 (Estimated); Status verified 2016-02

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Iguratimod; Methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Iguratimod monotherapy (Experimental)
  Interventions: Drug: Iguratimod
- Iguratimod and MTX combination (Experimental)
  Interventions: Drug: Iguratimod; Drug: Methotrexate
- MTX monotherapy (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Iguratimod — 25 mg/tablet, taken orally, 2 tablets/day (bid)
  Arms: Iguratimod and MTX combination; Iguratimod monotherapy
Drug: Methotrexate — 2.5 mg/tablet, taken orally once a week, 4 tablets/week (week 1-week 4) , 6 tablets/week (week 5- week 52)
  Arms: Iguratimod and MTX combination; MTX monotherapy

SUMMARY:
This study is intended to evaluate the efficacy and safety of Iguratimod alone or Iguratimod in combination with Methotrexate (MTX) versus Methotrexate alone in patients with Rheumatoid Arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of RA according to the diagnostic criteria of the American College of Rheumatology (ACR) (revised in 1987)
* Rheumatoid Arthritis for 3 months to 2 years from the time of the initial diagnosis
* Subjects have active RA at the time of screening
* Subjects are naive to MTX or RA related biologics
* Written informed consent

Exclusion Criteria:

* Preceding treatment with DMARDs, immunosuppressants (cyclophosphamide, cyclosporine, azathioprine, etc.), or Tripterygium within 4 weeks prior to study entry
* Chest x-ray abnormalities, such as tuberculosis, interstitial pulmonary fibrosis, etc.
* ALT >1.5×ULN, AST >1.5×ULN, Cr >135umol/L
* WBC<4×109/L，HGB<85g/L，PLT<100×109/L
* Subjects with serious cardiovascular, renal, hematologic or endocrine diseases
* Pregnant or lactating women
* Allergic to any of the study drugs
* History of alcoholism
* Subjects with mental illness
* Subjects receiving live vaccines recently
* Subjects participating in other clinical study within 3 months prior to study entry

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 910 (Actual)
Dates: Start 2012-05; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with ACR 20 response | week 52
Change from baseline in modified Total Sharp Score (mTSS) | week 52

SECONDARY OUTCOMES:
Change from baseline in mTSS | week 24
Percentage of patients achieving radiographic non-progression | week 24, week 52
Percentage of patients with ACR 20 response | week 12, week 24, week 40
Percentage of patients with ACR 50 response | week 12, week 24, week 40, week 52
Percentage of patients with ACR 70 response | week 12, week 24, week 40, week 52
Percentage of patients with Simplified Disease Activity Index (SDAI) ≤ 3.3 | week 12, week 24, week 40, week 52
Change from baseline in Health Assessment Questionnaire (HAQ) | week 12, week 24, week 40, week 52
Incidence of adverse events | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chunde Bao, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital Affiliated to Shanghai Jiaotong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Du F, Dai Q, Teng J, Lu L, Ye S, Ye P, Lin Z, Ding H, Dai M, Bao C; SMILE Group. The SMILE study: Study of long-term methotrexate and iguratimod combination therapy in early rheumatoid arthritis. Chin Med J (Engl). 2025 Jul 20;138(14):1705-1713. doi: 10.1097/CM9.0000000000003200. Epub 2024 Jul 26. PMID 39056160